CLINICAL TRIAL: NCT06442631
Title: An Individualized Video-based Stroke Education Platform for Stroke Survivors and Caregivers
Brief Title: MyStroke for Stroke Survivors and Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Christopher Favilla, Assistant Professor of Neurology at the University of Pennsylvania, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 850498
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Stroke, Acute; Ischemic Stroke, Acute
Keywords: stroke education; ischemic stroke; stroke knowledge
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Given the nature of the intervention (an educational platform), masking of participants is not feasible, but other key study members (and clinicians) will be blinded to the study assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard stroke education (No Intervention): Participants in this arm of the study will receive institutional standard stroke education during the course of the hospitalization, standardized across the 5 participating sites. Standard education consists of non-standardized verbal bedside education by the care team, a standardized stroke educational booklet, and standardized verbal instructions by the bedside nurse addressing stroke risk factors and medications.
- MyStroke + standard stroke education (Experimental): Participants in this arm of the study will receive institutional standard stroke education in addition to access to MyStroke, a personalized video-based education platform. Each participant will receive their personalized page via email or SMS, as per their preference, and they will receive automated nudges to visit educational material after hospital discharge.
  Interventions: Behavioral: MyStroke

INTERVENTIONS:
Behavioral: MyStroke — MyStroke is a video-based educational platform that curates brief educational videos to inform patients and caregivers about key aspects of their stroke. Upon registering a user, information regarding the patient's stroke etiology, relevant stroke risk factors, and stroke prevention medications are used to populate educational content that is relevant to the individual. Users receive automated nudges to revisit MyStroke after hospital discharge on day 1, 3, 5, 7, and weekly thereafter.
  Arms: MyStroke + standard stroke education

SUMMARY:
The goal of this multicenter randomized trial is to evaluate the impact of a personalized video-based stroke education platform on patient-centered and health system-centered outcomes. The main questions this study aims to address are:

1. Does a personalized, video-based educational platform improve stroke knowledge?
2. Does a personalized, video-based educational platform reduce post-discharge health system utilization?
3. Do different strategies of nudging improve engagement with educational material after hospital discharge?

In order to determine the effect of this personalized stroke education strategy, researchers will compare subjects who receive standard stroke education with those who receive the personalized stroke education platform in addition to standard standard education. Patient knowledge will be assessed 90-days after discharge. Study participants will include both stroke patients and caregivers, who will:

1. Receive standard education during the stroke hospitalization
2. Complete a survey on the day of hospital discharge to assess their baseline knowledge.
3. Half of the subjects will be randomly assigned to also receive access to the personalized stroke education platform on the day of discharge.
4. All subjects will complete two follow-up study visits (7 and 90 days after discharge) in order to complete surveys.

DETAILED DESCRIPTION:
Stroke education represents a unique opportunity to empower stroke survivors (and caregivers) to promote self-management, augment adherence, and reduce post-stroke healthcare utilization. Despite being a key quality metric for stroke centers, most patient and caregiver education is poorly retained and a common source of dissatisfaction. In fact, most survivors are unaware of the cause of their stroke, their modifiable risk factors, and how to properly respond to future stroke symptoms. Although there is no gold standard, most centers rely on a combination of bedside verbal communication and standardized printed materials. Prior work has clarified that effective and durable educational interventions benefit from engaging content, personalization, accessibility, and low cost/burden. Retention is very poor during the stroke hospitalization, but this can be overcome by promoting ongoing engagement after discharge.

To that end, our group developed a web-based educational platform (MyStroke) that leverages the electronic health record to personalize video-based educational content for each stroke survivor. Simple but engaging videos are curated to address each patient's stroke etiology, individualized risk factors, prescribed stroke prevention medications, and post-stroke lifestyle issues. This approach transforms point-of-care stroke education, and integrated nudges reveal opportunities for re-education and re-engagement after hospital discharge to achieve a durable impact. In a recent single-center pilot trial, MyStroke improved patient and caregiver satisfaction and improved key elements of stroke knowledge. The objective of this proposal is to build upon our encouraging preliminary experience and conduct a multicenter randomized trial to evaluate the impact of MyStroke on both patient-centered (stroke knowledge, self-efficacy, satisfaction, quality of life) and health system-centered outcomes (medication adherence and health system utilization).

Electronic nudges will leverage principles of behavioral economics (i.e. enhanced nudges) to promote ongoing engagement. Our preliminary data indicate that even bland nudges promote engagement, but here we propose to use both bland nudges and enhanced nudges, such that platform analytics will compare the influence of different nudge types. Use of technology in this context stands to bridge geographic distances, connect stakeholders, and increase access to information, but it important to recognize the potential to exacerbate inequities for elderly patients and those with limited access to technology. Issues of digital inclusivity will be evaluated to reveal opportunities for platform improvement. The MyStroke platform offers a scalable solution stroke education which imposes no burden on the clinical team due to its reliance on a limited number of input fields which can be harvested from the electronic health record to individualized content for each patient.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Admitted to hospital with clinical diagnosis of acute ischemic stroke (imaging confirmation not required)
* Stroke symptom onset within 30 days of enrollment
* Being discharged to either home or an acute rehabilitation facility
* Access to internet enabled device (smartphone, tablet, computer)
* Fluent in either English or Spanish (does not need to be native or primary language)
* Willingness and ability to sign informed consent

Exclusion Criteria:

* Severe aphasia (score of ≥2 on NIHSS item 9)
* Ischemic stroke that is attributed to a surgical procedure
* Resides in a skilled nursing facility prior to admission
* Being discharged to skilled nursing facility or long-term acute care facility
* Unwillingness or inability to participate in remote/virtual study visits
* A terminal or advanced condition that raises the possibility the subject may not survive 90 days
* Any other illness or condition that the investigator feels would pose a hazard to the subject from participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
The Stroke Patient Education Retention (SPER) survey | 90 days
  Total score from the 5-question SPER (scale 0-10; higher score reflects better knowledge)

SECONDARY OUTCOMES:
Patient satisfaction with stroke education | 90 days
  5-point Likert-scale (Q: I am satisfied with the quality of my stroke education; Answers range from strongly disagree to strongly agree)
Stroke etiology awareness | 90 days
  The proportion of patients who correctly identify their stroke etiology (multiple choice)
Stroke risk factor awareness | 90 days
  The proportion of patients who correctly identify at least one of their vascular risk factors (select all that apply)
Antithrombotic medication awareness | 90 days
  The proportion of patients who correctly identify all prescribed antithrombotic medications (free response)
Stroke Self-Efficacy Questionnaire (SSEQ) | 90 days
  Total score from the 13 item questionnaire (each item scored 0-10; total score 0-130; higher scores represent higher levels of self-efficacy)
EuroQoL EQ-5D-5L | 90 days
  A standardized measure of health-related quality of life across 5 domains. Each domain is scored using a 5-point ordinal scale (1-5), and the Level Sum Score (LSS) is calculated as the sum of the 5 scores (LSS range is 5-25, lower scores represent higher quality of life).
Medication adherence | 90 days
  This will be assessed based on pharmacy record review to quantify the Proportion of Days Covered (PDC). PDC is calculated by dividing the number of days with medications available by the total number of days in question (scored between 0 - 1; higher numbers represent more favorable adherence)
Emergency Department utilization | 90 days
  The number of Emergency Room visits will be summed in the first 90 days following hospital discharge
Urgent outpatient visits | 90 days
  The number of urgent outpatient visits with primary care and neurologist will be summed in the first 90 days following hospital discharge
Outpatient provider communication | 90 days
  The number of communications with primary care or neurology providers via telephone or provider communication apps will be summed in the first 90 days following hospital discharge

OTHER OUTCOMES:
The Stroke Patient Education Retention (SPER) survey (7 days) | 7 days
  Total score from the 5-question SPER (scale 0-10; higher score reflects better knowledge)
Patient satisfaction with stroke education (7 days) | 7 days
  5-point Likert-scale (Q: I am satisfied with the quality of my stroke education; Answers range from strongly disagree to strongly agree)
Stroke etiology awareness (7 days) | 7 days
  The proportion of patients who correctly identify their stroke etiology (multiple choice)
Stroke risk factor awareness (7 days) | 7 days
  The proportion of patients who correctly identify at least one of their vascular risk factors (select all that apply)
Antithrombotic medication awareness (7 days) | 7 days
  The proportion of patients who correctly identify all prescribed antithrombotic medications (free response)
Stroke Self-Efficacy Questionnaire (SSEQ) (7 days) | 7 days
  Total score from the 13 item questionnaire (each item scored 0-10; total score 0-130; higher scores represent higher levels of self-efficacy)
EuroQoL EQ-5D-5L (7 days) | 7 days
  A standardized measure of health-related quality of life across 5 domains. Each domain is scored using a 5-point ordinal scale (1-5), and the Level Sum Score (LSS) is calculated as the sum of the 5 scores (LSS range is 5-25, lower scores represent higher quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Favilla, MD, Principal Investigator — Assistant Professor of Neurology at the University of Pennsylvania
Locations (5):
- United States (5):
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Once a manuscript describing such data is accepted for publication, the deidentified dataset contributing to the publication will be shared publicly using the figshare repository (figshare.com). The availability of shared derived data will be described in publications and presentation.
Supporting Information: Study Protocol, SAP
Time Frame: We anticipate final sharing of data will take place at the completion of the 5-year project, but if an interim analysis results in a publication, the dataset will be shared at that time-point.
Access Criteria: The data will be publicly available and searchable on figshare (figshare.com), and the availability of shared derived data will be described in publications and presentation.